CLINICAL TRIAL: NCT01435915
Title: A Single Dose and Repeat Dose Study to Investigate the Pharmacokinetics of Ropinirole After Single and Multiple Doses of a PR-formulation in Chinese Healthy Male and Female Subjects
Brief Title: Ropinirole PR Pharmacokinetics Study Among Chinese Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 112558
Record Dates: First submitted 2011-09-01; First posted 2011-09-19 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — ropinirole

ARMS (1):
- Subjects receiving ropinirole (Experimental): Eligible subjects will receive single and multiple oral dose of ropinirole prolonged release tablet in sequence over 14 days without dosing on washout period from Day 2 to Day 7.
  Interventions: Drug: Ropinirole

INTERVENTIONS:
Drug: Ropinirole — Ropinirole 2 milligrams once daily prolonged release tablet will be given at 24-hour intervals in the morning.
  Single and repeat dose treatment periods will be separated by 7 days of washout period.

SUMMARY:
The purpose of this study is to investigate the pharmacokinetic profile of ropinirole PR after single and multiple doses of the PR-formulation. It will also investigate the safety and tolerability of ropinirole PR after single and multiple doses of PR-formulation.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult men and women between 18 and 45 years of age, inclusive.
2. Body weight >=50Kg.
3. Body Mass Index (BMI) 19 - 24 kg/m2.
4. No abnormality on clinical examination.
5. No abnormality revealed by the clinical chemistry or haematology examination at the pre-study medical examination.
6. A normal 12-lead ECG at the pre-study screening.
7. Normal systolic (100-140mmHg) and diastolic (<90mmHg) blood pressure at pre-study screening.
8. Written informed consent prior to admission to the study.

Exclusion Criteria:

1. Any clinically relevant abnormality identified on the screening history and physical or laboratory examination significant cardiovascular, neurological, psychiatric, haematological or renal abnormalities.
2. Definite or suspected personal history or family history of adverse reactions or hypersensitivity to the study drug or to drugs with a similar chemical structure.
3. History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
4. The subject has received prescribed medication within 7 days prior to the first dosing day, which in the opinion of the principal medical investigator interfered with the study procedures or compromised safety.
5. The subject has received over-the-counter (OTC) medicine within 48 hours prior to the first study day. Subjects who took OTC medication could still be entered into the study, if, in the opinion of the principal/co-investigator, the medication received did not interfere with the study procedures or compromised safety of the subjects.
6. Abuse of alcohol, defined as an average weekly intake of greater than 21 units or an average daily intake of greater than three units. One unit is equivalent to half a pint of beer, one measure of spirits or one glass of wine.
7. Positive screen for addictive drugs and tobacco.
8. Participation in a trial with any drug within the 1 month before the start of the study.
9. Either blood donation within the previous 3 months, or donation of a quantity of blood within the previous 12 months that would result in the subject having donated more than 1,500mL blood in a period from 12 months before this study up to and including the end of the study.
10. Positive pre-study screening result for hepatitis B antigen, hepatitis C antibody and HIV-1/2 antibodies.
11. Pregnancy and/or lactation;
12. Female subjects of childbearing potential who are intending to become pregnant and/or are not willing to avoid pregnancy by means of barrier contraception methods (i.e. condoms or IUD) during the study from 5 days prior to screening or in the 3 months following the study.
13. Female subjects with positive serum hCG test result at screening or on Days 1 of both study phases with positive urine HCG test.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-06-28 (Actual); Primary Completion 2010-08-05 (Actual); Study Completion 2010-08-05 (Actual)

PRIMARY OUTCOMES:
Profile of Pharmacokinetics | predose,1,2,3,4,6,8,10,12,14,16,18,20,22,24,36,48,72, 96,120,144,168 hours post-dose
  Cmax, AUC (0-24), AUC(0-inf)
Profile of Pharmacokinetics | predose,1,2,3,4,6,8,10,12,14,16,18,20,22,24 hours after last repeated dosing
  Css_max, Css_min and AUCss

SECONDARY OUTCOMES:
Profile of Pharmacokinetics | pre-dose,1,2,3,4,6,8,10,12,14,16,18,20,22, 24,36,48,72,96,120,144,168hours post-dose
  Tmax, T1/2, Kel
Composition of Pharmacokinetics | predose,1,2,3,4,6,8,10,12,14,16,18,20,22,24 hours after last repeated dosing
  Tmax, Css_av, DF，accumulation ratios (Ro and Rs)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Beijing, China

REFERENCES:
- See also: Results for study 112558 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/112558?search=study&study_ids=112558#rs